CLINICAL TRIAL: NCT00791089
Title: Effect of Omega-3 Fatty Acids on Short and Long-Term Maintenance of Sinus Rhythm After Radiofrequency Catheter Ablation for Atrial Fibrillation
Brief Title: Effects of Fish Oil on Post Ablation Arrhythmias
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: unable to secure funding and long term follow up
Sponsor: University of Michigan (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Hakan Oral, Cardiology EP Director, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LVZ111900
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-08

CONDITIONS: Atrial Fibrillation
Keywords: Radiofrequency Ablation; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Fish Oils; Omacor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fish Oil, Ablation, Sinus Rhythm (Experimental): Patients in the treatment arm will receive omega-3 fatty acids (EPA+DHA 4 gram/day) for 4 weeks before and 3 months after the ablation procedure.
  Interventions: Drug: LOVAZA Omega 3-acid ethyl esters; Drug: LOVAZA
- placebo, Ablation, sinus rhythm (Placebo Comparator): Patients in the control arm will not receive any omega-3 fatty acids. However they will receive placebo.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: LOVAZA Omega 3-acid ethyl esters — Treatment with omega-3 fatty acids (4g/day) for 4 weeks before and 3 months after radiofrequency catheter ablation for AF.
  Other Names: Fish Oil; Lovaza
  Arms: Fish Oil, Ablation, Sinus Rhythm
Drug: LOVAZA — (EPA+DHA 4 gram/day) for 4 weeks before and 3 months after the ablation procedure.
  Arms: Fish Oil, Ablation, Sinus Rhythm
Other: placebo — Control group will receive placebo before & after ablation.
  Arms: placebo, Ablation, sinus rhythm

SUMMARY:
To determine if peri-operative treatment with omega-3 fatty acids is associated with a decrease in the incidence of early recurrences of atrial arrhythmias (within 30 days) and an improvement in probability of long-term maintenance of sinus rhythm after radiofrequency catheter ablation for Atrial Fibrillation.

DETAILED DESCRIPTION:
AF is the most prevalent arrhythmia, affecting >2 million Americans. Antiarrhythmic drug therapy often is ineffective to eliminate recurrent episodes of AF. In recent years radiofrequency catheter ablation has emerged as a highly effective treatment strategy in patients with paroxysmal and chronic AF.6, 7 However, AF may recur within days to weeks after a successful ablation procedure in up to 50% of the patients, probably because of an inflammatory response to thermal injury caused by radiofrequency energy application. These early recurrences of AF after ablation do not necessarily predict long-term clinical outcome and 30-50% of patients who develop early recurrences ultimately remain in sinus rhythm without the need for additional ablation.8 However, early recurrences of AF may be associated with significant morbidity due to troubling symptoms of rapid ventricular rates, multiple hospital visits and cardioversions, need for antiarrhythmic drug therapy and prolongation in duration of anticoagulant therapy. It is also possible that if early recurrences of AF after ablation can be avoided, the probability of remaining in sinus rhythm during long-term follow-up may be higher, as maintenance of sinus rhythm early-on may facilitate reverse left atrial remodeling. A similar phenomenon may occur in post-operative AF, that develops in ~30% of patients who undergo cardiac surgery. Post-operative AF is often transient and usually resolves within 3 months after the surgery. Perioperative treatment with omega-3 fatty acids has been reported to decrease the incidence of postoperative AF after coronary artery by-pass surgery.4 Because the pathogenetic factors that play a role in postoperative AF and early recurrences of AF after radiofrequency catheter ablation may be similar, it is plausible that treatment with omega-3 fatty acids before and after ablation will be associated with a reduction in the incidence of early recurrences of AF.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 70 years old
* Left atrial size <55 mm

Exclusion Criteria:

* Inability or unwillingness to provide informed consent
* Current therapy with omega-3 fatty acids
* Current therapy with a statin
* Active liver disease
* Significant comorbidity such as end-stage renal disease or cirrhosis
* Valvular prosthesis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Oral, MD, Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Cardiovascular Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All of the 12 participants were assigned to an intervention, but none completed all aspects of the study, because of study termination due to funding withdrawal. Still, basic baseline and outcome measure data was available for 11 of the 12, as noted below.
Period: Overall Study
Arm/Group | Fish Oil, Ablation, Sinus Rhythm | Placebo, Ablation, Sinus Rhythm
Started | 6 | 6
Began Actually Taking Fish Oil or Placeb | 6 | 5
Six-month Data Collected | 6 | 5
Completed | 0 | 0
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Population: Baseline analysis is provided for all persons who actually began their assignment.
Groups:
- Fish Oil, Ablation: Patients in the treatment arm will receive omega-3 fatty acids (EPA+DHA 4 gram/day) for 4 weeks before and 3 months after the ablation procedure.
  LOVAZA Omega 3-acid ethyl esters: Treatment with omega-3 fatty acids (4g/day) for 4 weeks before and 3 months after radiofrequency catheter ablation for AF.
  LOVAZA: (EPA+DHA 4 gram/day) for 4 weeks before and 3 months after the ablation procedure.
- Total: Total of all reporting groups
Arm/Group | Fish Oil, Ablation | Placebo, Ablation, Sinus Rhythm | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Full Range); unit: years] — Population: One age for one participant randomized to this arm is unavailable. This participant actually never began placebo.
  years | 56 [43 to 64] | 48.8 [26 to 65] | 52.7 [26 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Normal Sinus Rhythm (Freedom From Atrial Arrhythmias)
Description: Freedom from atrial arrhythmias at 6 months will be defined as absence of any atrial arrhythmias with or without antiarrhythmic drug (AAD) therapy as shown in the two lines
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Placebo, Ablation: Patients in the control arm will not receive any omega-3 fatty acids. However they will receive placebo.
  placebo: Control group will receive placebo before & after ablation.
Arm/Group | Fish Oil, Ablation | Placebo, Ablation
Number analyzed (Participants) | 6 | 5
Participants
  FREEDOM FROM ATRIAL ARRHYTHMIAS WITHOUT AAD | 1 | 2
  FREEDOM FROM ATRIAL ARRHYTHMIAS WITH AAD | 3 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Fish Oil, Ablation | Placebo, Ablation
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fish Oil, Ablation (N=6) | Placebo, Ablation (N=6)
Cardiac Tamponnade (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fish Oil, Ablation (N=6) | Placebo, Ablation (N=6)
Anxiety (Psychiatric disorders) | 0 | 1
Fluid gain (Surgical and medical procedures) | 0 | 1
Spot on Face (Skin and subcutaneous tissue disorders) | 0 | 1
Painful vericose veins (Blood and lymphatic system disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
pneumonitis (Surgical and medical procedures) | 1 | 0

LIMITATIONS AND CAVEATS:
The Study was terminated before subject enrollment completion, due to financial concerns and loss of major support from the 21-day cardiac monitoring device. So small sample size means data should be interpreted with great caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes